CLINICAL TRIAL: NCT00750347
Title: Evaluation of the Interaction of Rimonabant (Antagonist of CB1 Receptor) on the Analgesic Effect of Paracetamol in Intravenous Administration
Brief Title: Antagonistic Interaction CB1-paracetamol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Pr Claude DUBRAY, CIC-CPC
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0037
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Pain
Keywords: pain,; analgesia; Healthy volunteers
MeSH Terms: conditions — Pain; Agnosia | interventions — Rimonabant; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Rimonabant and Paracetamol and placebo — evaluation of an possible inhibiting effect of rimonabant on the analgesic effect of paracetamol in healthy volunteers

SUMMARY:
Evaluation of an possible inhibiting effect of Rimonabant on the analgesic effect of Paracetamol in healthy volunteers

DETAILED DESCRIPTION:
Double Blind, cross-over, randomized and controlled versus placebo, study in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* between 18 and 40 years old
* written consent given

Exclusion Criteria:

* Rimonabant or paracetamol hypersensibility
* Excessive consumption of alcohol, tobacco, coffee, tea or toxicomania
* Concomitant medication
* Chronical diseases

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Pain's threshold with electrical stimulation (Pain Matcher). Pain's threshold with mechanical stimulation (electronical Von Frey). | during electrical stimulation

SECONDARY OUTCOMES:
Plasmatic concentration of paracetamol or his metabolite with or without Rimonabant | with or without rimonabant

CONTACTS AND LOCATIONS:
Overall Officials: Dubray Claude, Pr, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - CIC-CPC, Clermont-Ferrand
  - CHU Clermont-Ferrand, Clermont-Ferrand